CLINICAL TRIAL: NCT04727060
Title: A Prospective and Retrospective, Open Label Study to Collect Clinical Data to Document Clinical Performance and Safety in Total Knee Arthroplasty Using HLS Implants
Brief Title: Open Label Study to Collect Clinical Data to Document Clinical Performance and Safety in Total Knee Arthroplasty
Status: Terminated | Type: Observational
Why Stopped: the clinical data collected to date are sufficient for regulatory requirements
Sponsor: Corin (Industry)
Responsible Party: Sponsor
Other Study IDs: 0904-T-KNEE-RM
Record Dates: First submitted 2020-11-02; First posted 2021-01-27 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Total Knee Arthroplasty; Knee Disease; Total Knee Replacement; Osteo Arthritis Knee
Keywords: Knee Arthroplasty; Prosthesis; Implants; HLS implants; postero-stabilized prosthesis; third condyle; Arthroplasty
MeSH Terms: interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: patient with knee arthroplasty
  Other Names: patient with HLS prosthesis

SUMMARY:
The purpose of this study is to evaluate clinical performance and safety in total knee arthroplasty using HLS implants.

DETAILED DESCRIPTION:
It is planned to collect prospective and retrospective data from a continuous and exhaustive series of patients in a French center where Total Knee Arthroplasty with HLS prosthesis is performed routinely.

All patients treated with HLS KneeTec (cemented, non-cemented or hybrid versions) implant will be included. All eligible patients seen in consultation and who agree to participate in the study should be included, systematically and consecutively, since the initiation of the study.

Data will be collected retrospectively for HLS I, II, Evolution and Noetos® implants, and when prospectively for cementless, cemented and hybrid HLS KneeTec prosthesis.

Post-surgery visit data will be collected at 1-y , 3-y , 5-y, 10-y FU visits per protocol then up to the latest FU visit available.

ELIGIBILITY:
Inclusion Criteria:

* For the HLS-1, HLS-2, HLS Evolution and HLS Noetos retrospective group:

  1. Adult patients older than 18 years old.
  2. Patients who have undergone routine preoperative clinical evaluations prior to their Total Knee Replacement surgery and implanted with one of the following prostheses from the HLS range: HLS-1, HLS-2, HLS Evolution and HLS Noetos between their first date of use in 1987 and their last date of use as normal practice at the participating site in accordance to indications and intended use as described in the Instruction for Use (IFU) of the study devices.
  3. Patients who have been informed about their participation into an observational study.

For the HLS KneeTec prospective group (with retrospective surgeries):

1. Adult patients older than 18 years old.
2. Patients who have undergone routine preoperative clinical evaluations and received a TKR or are suitable candidates for a TKR with a fixed or mobile postero-stabilized HLS KneeTec prosthesis (cementless, cemented or hybrid combination) for the treatment of a primary or secondary knee osteoarthritis and inflammatory disease such as rheumatoid arthritis in accordance to indications and intended use as described in the Instruction for Use (IFU) of the study devices.
3. Patients who are willing and able to complete the scheduled FU visits.
4. Patients who have been informed about their participation into an observational registry study

Exclusion Criteria:

* Patients mentally incompetent or unable to understand what participation in the study entails.
* Patients who present signs and symptoms of any of the known contraindications described in the Instruction for Use (IFU) of the study devices.
* Patients who deny their participation into the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: It is planned to collect prospective and retrospective data from a continuous and exhaustive series of patients in a French center where Total Knee Arthroplasty with HLS prosthesis is performed routinely.
  All patients treated with HLS KneeTec (cemented, non-cemented or hybrid versions) implant will be included. All eligible patients seen in consultation and who agree to participate in the study should be included, systematically and consecutively, since the initiation of the study
Sampling Method: Non-Probability Sample
Enrollment: 2146 (Actual)
Dates: Start 2011-12-15 (Actual); Primary Completion 2023-11 (Actual); Study Completion 2023-11 (Actual)

PRIMARY OUTCOMES:
Evaluation of long-term survivorship of total knee replacement surgeries with HLS devices | 10-year
  Implants survival

SECONDARY OUTCOMES:
Evaluation of clinical performance | baseline (pre-surgery) to 10-year
  Change of clinical performance using the International Knee Society (IKS) score
Evaluation of patient satisfaction with the surgery | time up to 10-year FU
  Patients satisfaction post-surgery and any change during time up to 10-year FU using satisfaction questionnaire
Radiographic evaluation | baseline (1-year FU) to 10-year FU
  Implant positioning and stability, presence/absence of progressive radiolucent lines around implant components, any sign of loosening components via radiological evaluation from baseline (1-year FU) to 10-year FU.
Evaluation of safety of the study implants | time up to 10-year FU
  Number, severity and causal relationship of procedure or implant-related Adverse Events (AEs) starting intraoperatively up to 10-year FU.

CONTACTS AND LOCATIONS:
Overall Officials: Elvire SERVIEN, MD,PhD, Principal Investigator — Service de chirurgie orthopédique. Hopital de la Croix-Rousse, Hospices Civils de Lyon - France
Locations (1):
- Hopital de la Croix-Rousse, Hospices Civils de Lyon, Lyon, France